CLINICAL TRIAL: NCT00466921
Title: Phase II Trial of CC-5013 (Lenalidomide, Revlimid®) in Patients With Cutaneous T-Cell Lymphoma
Brief Title: Lenalidomide in Treating Patients With Relapsed Mycosis Fungoides/Sezary Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NU 04H5; P30CA060553 (NIH); NU-04H5
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Results first posted 2020-11-16 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-10

CONDITIONS: Lymphoma
Keywords: recurrent mycosis fungoides/Sezary syndrome; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome
MeSH Terms: conditions — Lymphoma; Mycosis Fungoides; Sezary Syndrome | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Lenalidomide (Experimental)
  Interventions: Drug: lenalidomide

INTERVENTIONS:
Drug: lenalidomide — 10 mg daily orally administered on days 1 - 21 followed by 7 days rest of a 28-day cycle, increasing dose by 5 mg every cycle, up to a maximum of 25 mg.

SUMMARY:
RATIONALE: Lenalidomide may stop the growth of mycosis fungoides/Sezary syndrome by blocking blood flow to the cancer.

PURPOSE: This phase II trial is studying how well lenalidomide works in treating patients with relapsed mycosis fungoides/Sezary syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the response rate and duration of response in patients with relapsed mycosis fungoides/Sézary syndrome treated with lenalidomide.
* Determine the progression-free survival of patients treated with this drug.

Secondary

* Determine the toxicity of this drug in these patients.
* Correlate the antiangiogenetic and costimulatory effects of this drug with clinical activity in skin biopsies from these patients.
* Assess the specific immune effector cell recruitment and augmentation of antitumor response in these patients. (Northwestern University only)

OUTLINE: This is a multicenter study.

Patients receive oral lenalidomide once daily on days 1-21. Treatment repeats every 28 days for 2 courses. Patients with progressive disease are removed from study. Patients achieving complete response receive 2 additional courses of treatment beyond complete response. Patients achieving partial response or stable disease may continue to receive lenalidomide as above for up to 2 years. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients undergo tissue biopsies at baseline and on day 1 of course 2. Tissue specimens are analyzed for vessel density, presence of adhesion molecules, and immunophenotyping of dermal infiltrate.*

NOTE: *At Northwestern University only, blood and tissue samples from 5-10 patients are collected. Peripheral blood samples are analyzed for immune cell repertoire (CD4+, CD8+ T cells, NK cells, NKT cells, CD4+, CD25+ T-regulatory cells, monocytes, and dendritic cell subsets), cell surface molecules, and for TH1/TH2-associated cytokines, such as interleukin (IL)-2, IL-4, IL-10, IL-12, interferon gamma, and tumor necrosis factor alpha, by flow cytometry at baseline, day 15 of course 1, and at the end of course 1. Immunological activation is assessed by analyzing surface expression of CD45RO and CTLA-4 on CD4+ and CD8+ T cells in blood and skin samples. Skin specimens are stored for future research studies on predictive markers of lenalidomide activity.

After completion of study treatment, patients are followed every 3 months for 1 year.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed mycosis fungoides/Sézary syndrome

  * Stage IA-IVB disease
* Must have failed ≥ 1 prior topical treatment, including any of the following:

  * Steroids
  * Nitrogen mustard
  * Retinoids
  * Phototherapy
  * Photochemotherapy
  * Radiotherapy
  * Total skin electron beam
* Measurable disease with ≥ 1 indicator lesion designated prior to study entry

  * Erythrodermic patients are eligible

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* WBC ≥ 3,000/mm³
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 2.2 mg/dL
* AST and ALT ≤ 2 times upper limit of normal
* Not pregnant or nursing
* Negative pregnancy test
* Fertile women must use effective double-method contraception for ≥ 4 weeks before, during, and for ≥ 4 weeks after completion of study therapy
* Fertile men must use effective contraception during and for ≥ 4 weeks after completion of study therapy
* No other malignancy within the past 5 years except treated squamous cell and basal cell carcinoma of the skin, carcinoma in situ of the cervix, or surgically removed melanoma in situ of the skin (stage 0), with histologically confirmed free margins of excision and no current evidence of disease
* No acute infection requiring systemic treatment
* No known allergic reaction or hypersensitivity to thalidomide

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* More than 4 weeks since prior topical therapy, systemic chemotherapy, or biological therapy
* No prior stem cell transplantation
* No other concurrent systemic antipsoriatic or anticancer therapies, including radiotherapy, thalidomide, or other investigational agents
* No other concurrent topical agents except emollients

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2005-04-19 (Actual); Primary Completion 2010-04-05 (Actual); Study Completion 2013-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy M. Kuzel, MD, Study Chair — Robert H. Lurie Cancer Center
Locations (3):
- United States (3):
  - Stanford Cancer Center, Stanford, California
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas

REFERENCES:
- [Derived] Querfeld C, Rosen ST, Guitart J, Duvic M, Kim YH, Dusza SW, Kuzel TM. Results of an open-label multicenter phase 2 trial of lenalidomide monotherapy in refractory mycosis fungoides and Sezary syndrome. Blood. 2014 Feb 20;123(8):1159-66. doi: 10.1182/blood-2013-09-525915. Epub 2013 Dec 11. PMID 24335103

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened February 24, 2004 to accrual with the first patient being treated on study April 19 2005. the study closed to further accrual February 7, 2011 after the last patient initiated study treatment.
Groups:
- Lenalidomide: lenalidomide: 25 mg daily orally administered on days 1 - 21 followed by 7 days rest of a 28-day cycle, or starting dose of 10mg increasing dose by 5 mg every cycle, up to a maximum of 25 mg.
Period: First 3 Cycles of Treatment
Arm/Group | Lenalidomide
Started | 33 (One patient completed only a few days of treatment)
Completed 1 Cycle | 32
Started Cycle 2 | 31
Completed 3 Cycles | 26
Completed | 26
Not Completed | 7
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 5
Period: Completed 4 Cycles/Reached 1st Response
Arm/Group | Lenalidomide
Started | 26
Completed 4 Cycles/1st Response | 21
Completed | 21
Not Completed | 5
Not completed — Withdrawal by Subject | 2
Not completed — Progressive Disease | 2
Not completed — Other | 1
Period: Continued Treatment
Arm/Group | Lenalidomide
Started (Patients with partial response/stable disease continued for up to 2 years of treatment. Patients with complete response were treated with up to 2 more cycles.) | 21
Completed | 21
Not Completed | 0
Period: Follow up for a Minimum of 1 Year
Arm/Group | Lenalidomide
Started (All patients who have at least one dose of study treatment go into follow up for survival endpoints.) | 33
Completed | 27
Not Completed | 6
Not completed — Death | 6

BASELINE CHARACTERISTICS:
Arm/Group | Lenalidomide
Number analyzed (Participants) | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 6
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 33

OUTCOME MEASURES:

1. Primary Outcome: Response to Treatment
Description: In general response to treatment is defined as either complete response (CR) or partial response (PR) assessed using Composite Assessment (CA) of index lesion disease severity and is defined as the following:
  CR =CA ratio=0/no evidence of new disease (abnormal or pathologically positive lymph nodes, cutaneous or other tumor manifestations, visceral disease) present over 4 weeks. Patients with Sézary Syndrome must have no evidence of circulating Sézary cells (< 5% Sézary cells=not significant). Skin biopsy is required for documentation of CR. Confirmatory CT scans are required, if baseline CTs were abnormal.
  PR= CA ratio ≥0.5/no new clinically abnormal lymph nodes/no progression of existing clinically abnormal lymph nodes (<25%)/no new cutaneous tumors/no new pathologically positive lymph nodes or visceral disease in an area previously documented as-ve for at least 4 weeks. In patients with circulating Sézary cells at least a 50% reduction of malignant lymphocytes is required.
Time Frame: After cycle 4 of treatment (1 cycle =28 days)
Population: Patients considered not evaluable if they did not complete 1 cycle or were not evaluated for response
Measure: Number; unit: participants
Arm/Group | Lenalidomide
Number analyzed (Participants) | 29
participants
  CR | 0
  PR | 9

2. Primary Outcome: Progression-free Survival (PFS)
Description: PFS is defined from the time of treatment initiation until documentation of progressive disease or death from any cause.
  Progressive disease is defined as (PD) ≥25% increase in CA ratio, ≥25% increase in no. or area of clinically abnormal lymph nodes/new tumors/new pathologically positive lymph nodes/visceral disease/an increase >25% in no. of Sézary cells.
Time Frame: From time of treatment initiation until progression or death from any cause (up to a possible maximum of approximately 6 years)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 32
months | 8 [3.7 to 26.1]

3. Primary Outcome: Duration of Response (DOR)
Description: DOR is defined as time of initial documentation of response to the time of documentation of progression in patients who achieve either a complete response (CR) and partial response (PR)
Time Frame: From time of initial response until progressive disease (up to approximately 1 year)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Lenalidomide
Number analyzed (Participants) | 9
months | 10 [1.1 to 11.0]

4. Secondary Outcome: Number of Patients Who Experience Toxicity as Assessed by NCI CTCAE v3.0
Description: Toxicity is defined as the number of patients who patients who experienced an adverse event that was determined to be at least possibly related to study drug and determined to be a grade 3 or higher in severity as assessed by the Common Terminology Criteria for Adverse Events v3.0 (CTCAE) where generally:
  Grade 1 Mild AE Grade 2 Moderate AE Grade 3 Severe AE Grade 4 Life-threatening or disabling AE Grade 5 Death related to AE
Time Frame: From treatment initiation until up to 30 days post treatment with possible 4 cycles of initial treatment (1 cycle =28 days) and up to 2 further years of treatment permitted if meeting response criteria
Measure: Number; unit: patients
Arm/Group | Lenalidomide
Number analyzed (Participants) | 33
patients
  Fatigue (grade 3) | 7
  Infection (grade 3) | 1
  Leukopenia (grade 3) | 1

5. Other Pre Specified Outcome: Specific Immune Effector Cell Recruitment and Augmentation of Antitumor Response at Baseline and Day 15 of Course 1 (Northwestern University Only)
Time Frame: After all patients have completed thru day 15 of course 1.
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Correlation of Antiangiogenetic and Costimulatory Effects With Clinical Activity at Baseline and After Course 1
Time Frame: After all patients have completed 1 course
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Patients were assessed for adverse events from the time of treatment initiation until treatment discontinuation and up to 30 days post last treatment. Patients received a possible 4 cycles of initial treatment (1 cycle =28 days) and up to 2 further years of permitted treatment if meeting response criteria.
Arm/Group | Lenalidomide
All-Cause Mortality (participants affected / at risk) | 18/33
Serious Adverse Events (participants affected / at risk) | 10/33
Other Adverse Events (participants affected / at risk) | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=33)
Pneumonia (Infections and infestations) | 1
Pogression of disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Infection (Infections and infestations) | 2
Death more than 30 days from last dose of study drug (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Death dues to acute disseminated encephalomielitis (Nervous system disorders) | 1
Edema (Blood and lymphatic system disorders) | 1
Mental Status Changes (PVD) (Nervous system disorders) | 1
Leg infection (cellulitis) (Infections and infestations) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Lenalidomide (N=33)
Allergic rhinitis (including sneezing,nasal stuffiness,postnasal drip) (General disorders) | 1
Hemoglobin (anemia) (Blood and lymphatic system disorders) | 14
Neutrophils (neutropenia) (Blood and lymphatic system disorders) | 4
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 9
Increased white blood cells (Blood and lymphatic system disorders) | 1
Platelets (thrombocytopenia) (Blood and lymphatic system disorders) | 5
Hypotension (Cardiac disorders) | 2
Fatigue (General disorders) | 23
Fever (General disorders) | 1
Chills (General disorders) | 6
Sweating (General disorders) | 2
Weight loss (General disorders) | 2
Insomnia (General disorders) | 1
Cold intolerance (General disorders) | 1
Weight gain (General disorders) | 2
Injection site reaction/extravasation changes (Skin and subcutaneous tissue disorders) | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 19
erythoderma (Skin and subcutaneous tissue disorders) | 3
Rash (Skin and subcutaneous tissue disorders) | 4
Burning (Skin and subcutaneous tissue disorders) | 3
Skin peeling (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1
Scaling (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Hot flashes/flushes (Endocrine disorders) | 1
Thyroid function, high (hyperthyroidism) (Endocrine disorders) | 1
Anorexia (Gastrointestinal disorders) | 4
Constipation (Gastrointestinal disorders) | 7
Diarrhea (Gastrointestinal disorders) | 9
Heartburn/dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
dry mouth (Gastrointestinal disorders) | 1
Taste alteration(dysgeusia) (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Dysphagia (difficulty swallowing) (Gastrointestinal disorders) | 1
Inflammatory bowel disease (Gastrointestinal disorders) | 1
Abdominal bloating (Gastrointestinal disorders) | 1
Lung (pneumonia) (Infections and infestations) | 2
Infection (NOS) (Infections and infestations) | 8
Edema (Blood and lymphatic system disorders) | 5
Edema extremities (Blood and lymphatic system disorders) | 13
Alkaline phosphatase (Metabolism and nutrition disorders) | 2
Transaminase (Metabolism and nutrition disorders) | 5
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 10
Bilirubin (hyperbilirubinemia) (Metabolism and nutrition disorders) | 2
Creatinine Increased (Metabolism and nutrition disorders) | 3
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 1
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 4
Potassium, serum-low(hypokalemia) (Metabolism and nutrition disorders) | 1
Neurosensory (Nervous system disorders) | 5
Neuromotor (Nervous system disorders) | 1
Slurred speech (Nervous system disorders) | 1
Speech impairment (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Confusion (Nervous system disorders) | 1
Dizziness (Psychiatric disorders) | 2
Mood alteration - Depression (Psychiatric disorders) | 4
Muscle aches (Musculoskeletal and connective tissue disorders) | 1
Muscle cramps (Musculoskeletal and connective tissue disorders) | 3
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 2
Joint aches (Musculoskeletal and connective tissue disorders) | 1
muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
GENERAL- Pain (General disorders) | 12
Back pain (Musculoskeletal and connective tissue disorders) | 1
Pain in hands (Musculoskeletal and connective tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnea on exertion (Respiratory, thoracic and mediastinal disorders) | 1
Visual (Eye disorders) | 1
Renal insufficiency (Renal and urinary disorders) | 1
fratured coccyx (Injury, poisoning and procedural complications) | 1
Tumor flare - skin lesions (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
hypothyroid (Endocrine disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No